CLINICAL TRIAL: NCT00921531
Title: Phase Ⅲ Study of Adjuvant Therapy With Thalidomide for Chemoembolization in Advanced Hepatocellular Carcinoma
Brief Title: Adjuvant Therapy With Thalidomide for Chemoembolization in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: ethic committee of Zhongshan Hospital of Fudan University, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI-THALIDOMIDE; LCI-09-06-15
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2009-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; thalidomide; TACE; Child-Pugh Class A or B
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide and TACE (Experimental): Thalidomide is used for adjuvant therapy for TACE
  Interventions: Drug: Thalidomide; Drug: TACE
- TACE only (Active Comparator)
  Interventions: Drug: TACE

INTERVENTIONS:
Drug: Thalidomide — Thalidomide is used for adjuvant therapy for TACE
  Thalidomide will be given at the dose of 200 mg/day in beginning, with dose escalation of 100 mg/day each week, until to the dosage of 400 mg/day.
  Arms: Thalidomide and TACE
Drug: TACE — TACE (5-FU 1.0 g, OXP 150mg, MMC 10 mg, lipiodol 5-30 ml) will be performed every two months (defined as a course) until no radiological evidence of survival of tumor (based on contrast MRI) or 6 courses.

SUMMARY:
Chemoembolization (TACE) is used in the majority of advanced hepatocellular carcinomas. Randomized clinical trials indicated that TACE improves overall survival in patients with good liver function (Child-pugh A or B). However, the shortcoming of TACE is obvious: hypoxia induced neoangiogenesis after blockage of blood supply of the tumor; repeat TACE deteriorates liver cirrhosis due to toxicity of chemotherapeutic agent to the parenchyma liver. Thalidomide has been reported to have antiangiogenic and antimetastatic effects. The objectives of adjuvant therapy with thalidomide for chemoembolization is to evaluate overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma confirmed with pathology or identified with radiological images with typical features
* Age ≥ 18 years and ≤ 80 years
* At least one tumor nodule with one uni-dimension of ≥ 2 cm
* Child-Pugh Class A or B
* Total bilirubin ≤ 1.5 x upper limit of normal
* ALT and AST ≤ 2.0 x the upper limit of normal
* PT-INR<2.3,PTT < 1.5 x upper limit of normal
* Serum creatinine ≤ 1.5x upper limit of normal
* Peripheral white blood cell count of or more than 3×10(9)/L
* Peripheral platelet of or more than 50×10(9)/L
* Expected survival time not less than 3 months
* ECOG score 0-2

Exclusion Criteria:

* Tumor thrombi in main branch of portal vein
* Tumor involvement more than 70% of whole liver
* With extrahepatic metastasis
* Prior systemic chemotherapy or chemoembolization
* Congestive heart failure > NYHA class 2
* History of HIV infection
* Active clinically serious infections (> 2 NCI-CTC Version 3.0)
* Recurrence of HCC after liver transplantation
* Pregnant or breast-feeding
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in this study
* Known or suspected allergy to any agent given in association with this trial
* Patients unable to swallow oral medication
* Inclined to thrombosis
* Inclined to hemorrhage or active hemorrhage with 1 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months
  primary outcome is defined as overall survival. overall survival is calculated from the time of undergo treatment (TACE) to time of patients death.

SECONDARY OUTCOMES:
time to progression | 36 months
  time to progression is defined as from the time of treatment (TACE) to the time of patient's progression. the progression is defined as disease progression based on RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Cancer Institute, Shanghai, Shanghai Municipality, China

REFERENCES:
- See also: Fudan University,Shanghai,China — http://www.fudan.edu.cn/